CLINICAL TRIAL: NCT03002701
Title: The Impact of nUrsiNg DEliRium Preventive INterventions in the Intensive Care Unit (UNDERPIN-ICU): A Multi-centre, Stepped Wedge Randomized Controlled Trial
Brief Title: The Impact of Nursing Delirium Preventive Interventions in the Intensive Care Unit
Acronym: UNDERPIN-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UNDERPIN-ICU
Record Dates: First submitted 2016-11-25; First posted 2016-12-26 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Delirium
Keywords: Prevention; Critical care; Delirium; Nurse; RCT
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control - standard care (No Intervention): Prior to implementation of the intervention package the current standard of care will be maintained.
- Intervention group (Active Comparator): After implementation the intervention package will be implemented as standard care.
  Interventions: Behavioral: UNDERPIN-ICU program

INTERVENTIONS:
Behavioral: UNDERPIN-ICU program — UNDERPIN-ICU consists of standardized protocols focusing on several modifiable risk factors for delirium, including cognitive impairment, sleep deprivation, immobility and visual and hearing impairment.
  Arms: Intervention group

SUMMARY:
Delirium is a common disorder in Intensive Care Unit (ICU) patients and is associated with serious short- and long-term consequences. This study focuses on a program of standardized nursing and physical therapy interventions to prevent delirium in the ICU, and determines the effect of the program on the number of delirium-coma-free days in 28 days and several secondary outcomes in a multicenter randomized controlled trial.

DETAILED DESCRIPTION:
Delirium is a common disorder in Intensive Care Unit (ICU) patients and is associated with serious short- and long-term consequences, including re-intubations, ICU readmissions, prolonged ICU and hospital stay, persistent cognitive problems, and higher mortality rates. Considering the high incidence of delirium and its consequences, prevention of delirium is imperative. This study focuses on a program of standardized nursing and physical therapy interventions to prevent delirium in the ICU, called UNDERPIN-ICU (nUrsiNg DEliRium Preventive INterventions in the ICU).

Objective: To determine the effect of the UNDERPIN-ICU program on the number of delirium-coma-free days in 28 days and several secondary outcomes, such as delirium incidence, the number of days of survival in 28 and 90 days and delirium-related outcomes.

Design and Setting: A multicenter stepped wedge cluster randomized controlled trial.

Methods: Eight to ten Dutch ICUs will implement the UNDERPIN-ICU program in a randomized order. Every two months the UNDERPIN-ICU program will be implemented in an additional ICU following a two months period of staff training. UNDERPIN-ICU consists of standardized protocols focusing on several modifiable risk factors for delirium, including cognitive impairment, sleep deprivation, immobility and visual and hearing impairment.

Participants: ICU patients aged ≥ 18 years (surgical, medical, or trauma) and at high risk for delirium, E-PRE-DELIRIC ≥35%, will be included, unless delirium was detected prior ICU admission, expected length of ICU stay is less then one day or when delirium assessment is not possible.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years
* surgical, medical or trauma patients
* admitted to one of the participating ICUs
* at high risk for delirium (>35% determined with the E-PRE-DELIRIC prediction tool)

Exclusion Criteria:

* delirious before ICU admission
* an ICU stay < one day
* reliable assessment for delirium is not possible due to: sustained coma; serious auditory or visual disorders; inability to understand Dutch; severely mentally disabled; serious receptive aphasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1750 (Actual)
Dates: Start 2016-12-31 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
The number of delirium-coma-free days | 28 days
  The number of days a patient is not delirious and not in coma in 28 days starting from the day of inclusion in the study after ICU admission.

SECONDARY OUTCOMES:
Delirium incidence | 28 days
  One or more episodes of positive delirium screening after ICU admission.
The number of days of survival | 28 days
  The number of days survived since ICU admission.
The number of days of survival | 90 days
  The number of days survived since ICU admission.
Duration of mechanical ventilation | 28 days
  The number of days a patient was mechanically ventilated.
Incidence of re-intubation | 28 days
  Patients who need to be intubated within 28 days after ICU admission, following a previous extubation, irrespectively the reason for re-intubation, will be counted as incident case for re-intubation.
Incidence of ICU re-admission | 28 days
  Patients who need to be readmitted to the ICU within 28 days, irrespectively the reason for readmission, will be counted as incident cases for ICU readmission.
Incidence of unplanned removal of tubes/catheters | 28 days
  Incidents in which patients remove their tube or catheter themselves will be counted as incident cases for unplanned removal. The period in which this is measured is during patients' ICU stay or during the period when the patient is delirious (in case a patient is discharged to the ward) with a maximum of 28 days.
Incidence of physical restraints | 28 days
  Patients who need physical restraints (fixation of their limbs to prevent them from removing tubes or lines) within 28 days, will be counted as incident cases for physical restraints.
ICU length of stay | 365 days
  This is defined as the number of days a patient is admitted to the ICU. Hospital length of stay is defined as number of days a patient is admitted to the hospital.
Hospital length of stay | 365 days
  This is defined as the number of days a patient is admitted to the ICU. Hospital length of stay is defined as number of days a patient is admitted to the hospital.
Health related quality of Life (HRQoL) | 90 days after ICU admission
Health related quality of Life (HRQoL) | 365 days after ICU admission
Post-hoc analysis | During admission
Cost-effectiveness | During ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Mark van den Boogaard, PhD, Principal Investigator — Radboud University Medical Center
Locations (11):
- Netherlands (11):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Hospital Gelderse Vallei, Ede
  - Medical Spectrum Twente, Enschede
  - Hospital St. Jansdal, Harderwijk
  - Medical Center Leeuwarden, Leeuwarden
  - Haaglanden Medical Center location Westeinde, The Hague
  - Hospital ETZ location Elisabeth, Tilburg
  - Hospital ETZ location Tweesteden, Tilburg
  - Bernhoven Hospital, Uden
  - Maxima Medical Center, Veldhoven
  - ISALA clinics, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wassenaar A, Rood P, Schoonhoven L, Teerenstra S, Zegers M, Pickkers P, van den Boogaard M. The impact of nUrsiNg DEliRium Preventive INnterventions in the Intensive Care Unit (UNDERPIN-ICU): A study protocol for a multi-centre, stepped wedge randomized controlled trial. Int J Nurs Stud. 2017 Mar;68:1-8. doi: 10.1016/j.ijnurstu.2016.11.018. Epub 2016 Dec 8. PMID 28013104
- [Derived] Tilburgs B, Rood PJT, Zegers M, van den Boogaard M; UNDERPIN-ICU study group. The implementation of nUrsiNg DEliRium preventive INterventions in the Intensive Care Unit (UNDERPIN-ICU): A qualitative evaluation. Int J Nurs Stud. 2023 Jan;137:104386. doi: 10.1016/j.ijnurstu.2022.104386. Epub 2022 Nov 8. PMID 36427481
- [Derived] Rood PJT, Zegers M, Ramnarain D, Koopmans M, Klarenbeek T, Ewalds E, van der Steen MS, Oldenbeuving AW, Kuiper MA, Teerenstra S, Adang E, van Loon LM, Wassenaar A, Vermeulen H, Pickkers P, van den Boogaard M; UNDERPIN-ICU Study Investigators. The Impact of Nursing Delirium Preventive Interventions in the ICU: A Multicenter Cluster-randomized Controlled Clinical Trial. Am J Respir Crit Care Med. 2021 Sep 15;204(6):682-691. doi: 10.1164/rccm.202101-0082OC. PMID 34170798
- See also: Related Info — http://dx.doi.org/10.1016/j.ijnurstu.2016.11.018